CLINICAL TRIAL: NCT00993538
Title: Leukemia Cell Cultures for Research of New Anti-cancer Therapies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER/Directeur de la Recherche Clinique et des Innovations, University Hospital, Strasbourg, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4452
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Acute Leukaemia
Keywords: Leukaemia; Blood and marrow cells culture; Cell growth; Cell differentiation
MeSH Terms: conditions — Leukemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Blood sampling; Procedure: Bone marrow aspiration

INTERVENTIONS:
Procedure: Blood sampling
Procedure: Bone marrow aspiration

SUMMARY:
The main objective of this project is not only a better understanding of the human leukemic disease but also to find new anti-leukemic or improve existing ones. This study has, the following aims:

* To analyze the genetic and epigenetic regulation of the retinoic acid induced cascade which leads to the expression of TRAIL in blood cells of patients with acute leukemia. This study will be complemented by the analysis of global gene expression (DNA chips) and of the DNA methylation state, and by chromatin immunoprecipitation experiences.
* To determine the efficiency of inhibitors of enzymes responsible for the modification of chromatin (existing and new developments within the European consortium EPITRON coordinated by Dr Gronemeyer) as inducers of differentiation and / or apoptosis of leukemic blasts.
* To explore Ikaros genic and functional abnormalities (genomic deletions, mutations, abnormal transcripts and proteins) in acute leukemia. The aim is to determine if these abnormalities may play a prognosis role.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected de novo or secondary or relapsed acute leukemia, requiring complementary blood test and bone marrow analysis
* Patients older or equal than 28 days
* Informed consent signed

Exclusion Criteria:

* Pregnancy
* Breastfeeding

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-07

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Herbrecht, MD, Principal Investigator — Département d'Hématologie et d'Oncologie-hôpital de Hautepierre Strasbourg, France
Locations (2):
- France (2):
  - Service d'Hématologie et d'Oncologie, Strasbourg
  - Service de Pédiaterie - Hôpital de Hautepierre, Strasbourg